CLINICAL TRIAL: NCT00414024
Title: An Open Label 52-week Study to Evaluate the Safety and Efficacy of Tegaserod Given Orally for the Treatment of Opioid-induced Constipation (OIC) in Patients With Chronic Non-cancer Pain
Brief Title: Safety and Efficacy of Tegaserod in Opioid-induced Constipation in Patients With Non-cancer Pain.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early as a result of regulatory action suspending tegaserod use in 2007
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHTF919N2302
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Opioid-induced Constipation
Keywords: Opioid, constipation, tegaserod
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study will evaluate the safety and efficacy of Tegaserod in opioid-induced constipation in patients with non-cancer pain.

Patients who enter this study PRIOR to the core study (CHTF919N2201) interim analysis receive the treatment as follows:

Patients will be randomly assigned to receive open label tegaserod 6 mg b.i.d. or tegaserod 12 mg o.d. using an allocation ratio of 1:1.

Patients who enter this study AFTER the core study interim analysis receive the treatment as follows:

Patients will be assigned to receive the selected tegaserod dose regimen (as determined by the core study interim analysis) in an open label fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 years of age or older.
* Patients with chronic non-cancer pain that necessitates the use of non- injectable opioid analgesics.
* Chronic pain which has been present for a minimum of 3 months which needs the chronic use of opioids for pain relief.
* Constipation, according to the investigator's clinical judgment, that is resulting from opioid use for non-cancer chronic pain. Opioid-induced Constipation (OIC) is defined as follows:

less than 3 spontaneous bowel movements per week and at least one of the following on at least 25% of occasions:

1. Hard or very hard stools
2. sensation of incomplete evacuation
3. straining while having a bowel movement

Exclusion Criteria:

* 1. Who are receiving opioids for abdominal pain or connective tissue disorders.
* Planned discontinuation of opioids during the study
* Who underwent major surgery within 3 months prior to screening.
* With a history of prior chronic constipation (CC) that was present for more than three months and that was not related to opioid use.
* With a current diagnosis of irritable bowel syndrome (IBS) constipation predominant or alternators.
* With a previous use of tegaserod within 3 months prior to baseline.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the long term safety of tegaserod

SECONDARY OUTCOMES:
Change from baseline assessment of OIC symptoms at weeks 24 and 52
Change from baseline assessment of opioid-induced mid/upper GI symptoms at weeks 24 and 52
Patients weekly assessment of intensity of pain for which opioids were prescribed at weeks 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corp., Principal Investigator — NPC
Locations (6):
- 60 Investigative Sites, East Hanover, New Jersey, United States
- 2 Investigative Sites, Hong Kong, China
- 6 Investigative Sites, Egypt, Egypt
- 1 Investigative Site, Singapore, Singapore
- 2 Investigative Sites, Dawan, Taiwan
- 4 Investigative Sites, Venezuela, Venezuela